CLINICAL TRIAL: NCT04356924
Title: Evaluation of a Novel Psychological Intervention Tailored for Patients With Early Cognitive Impairment (PIPCI)
Brief Title: Psychological Treatment to Support the Consequences of Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Urban Ekman, Assistant Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KIPT6692021
Record Dates: First submitted 2020-04-15; First posted 2020-04-22 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Cognitive Impairment; Psychological; Psychotherapy; Health Behavior
Keywords: Cognitive impairment; Psychological treatment; Dementia prevention
MeSH Terms: conditions — Cognitive Dysfunction; Health Behavior | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Psychological treatment (Experimental): The psychological treatment consists of 11 sessions (55 minutes per occasion), where the patient meets a psychologist face-to-face (either licensed or under training to be licensed) once a week. In between sessions, patients are supposed to complete homework exercises that are related to the contiguous sessions (2 x 45 minutes per week).
  Interventions: Behavioral: Psychological treatment
- Cognitive training (Active Comparator): Like the experimental group, the active control group also consists of 11 sessions (55 minutes per occasion), once a week. At those occasions, the patient will meet a psychology student under training or a MSc in psychology that coaches the patients during the cognitive training. In between sessions, patients are supposed to take 2 walks (45 minutes per occasion to meaningfully match the home exercises in the experimental group).
  Interventions: Behavioral: Cognitive training
- Treatment as usual (No Intervention): This group receives no intervention. They receive regular health information that is given after the extended cognitive examination at the Cognitive Centers. However, after the finalization of the post-intervention evaluations, this group will be randomized to participate in one of the active interventions. We will conduct additional post-intervention assessments also for those individuals in this group that accept this offer to increase the power of the intervention evaluation.

INTERVENTIONS:
Behavioral: Psychological treatment — The treatment is an adjusted (to the cognitively impaired individual) combination of CBT, ACT, validation strategies, and psychoeducation. One focus is to increase motivation to lifestyle changes, and to a larger degree live life in correspondence with internal goals.
  Arms: Psychological treatment
Behavioral: Cognitive training — Computer based training tasks implemented with adaptive intensity. The cognitive training method that will be used is mainly related to executive control (i.e., ability to coordinate thoughts and actions in accordance with internal goals).
  Arms: Cognitive training

SUMMARY:
The burden of cognitive impairment is severe, and often hinders affected people to act independently in daily life. Individuals in different stages of cognitive decline are frequently affected by existential distress and associated health issues (such as stress symptoms, anxiety, and depression), as well as social avoidance due to the unclear prognosis. Although the need for psychological support is large, there is a lack of efficient individualized psychological treatments- and methods to maintain psychological health that sufficiently impact daily life and promote behavioral- and biological change. In keeping with that notion, the investigators have developed a novel psychological treatment manual focused on supporting individuals with early phase cognitive impairment. The treatment manual is centered on facilitating behavioral change in accordance with personal values and long-term goals even in the presence of negative experiences, as well as to promote meaningful life-style changes. Conceptually, the treatment manual has its basis in the cognitive behavioral therapy (CBT) tradition, but the investigators have strived to adapt the manual to suit a cognitively affected population. The investigators will evaluate the psychological treatment in a RCT were the investigators will include approximately 138 individuals in their early phases of cognitive decline and randomize them into either an experimental group (psychological treatment), an active control group (cognitive training), or a treatment as usual control group. Evaluations will be conducted with, psychological health measures, cognitive assessments, and with biological markers.

The investigators hypothesize that in comparison with the control conditions, the response to psychological treatment will be associated with improved psychological health and improved cellular protection.

DETAILED DESCRIPTION:
Background

The burden of cognitive impairment is severe, and often hinders affected people to act independently in daily life, and their families frequently carry a large burden. A great challenge is to support the maintenance of cognitive health in order to avoid cognitive disability. Individuals diagnosed with subjective cognitive decline (SCD [unimpaired performance on cognitive tests]), mild cognitive impairment (MCI [Impaired performance on cognitive tests]) are frequently affected by health issues (such as stress symptoms, anxiety, and depression), as well as social avoidance due to the unclear prognosis of their cognitive dysfunction. Thus, the need for efficient psycho-social support are utterly needed both from an individual- as well as a societal perspective.

The investigators have developed a novel psychological treatment manual focused on supporting individuals with SCD and MCI. The treatment manual is centered on facilitating behavioral change in accordance with personal values and long-term goals even in the presence of negative experiences, as well as to promote meaningful life-style changes. The treatment manual has its basis in the cognitive behavioral therapy (CBT) tradition, but the investigators have strived to adapt the manual to suit a cognitively affected population with for example with reminders, more sessions, validation techniques, repetition, and concrete examples etc. Recent developments within CBT, particularly acceptance commitment therapy (ACT), emphasize the utility of acceptance and mindfulness strategies, contrasting interventions focused on reduction or control of symptoms. In brief, the treatment objective in ACT and in our study is to improve functioning by increasing psychological flexibility. Psychological flexibility is defined as the ability to notice and accept interfering thoughts, emotions and bodily sensations without acting on them, to facilitate behaving in accordance with personal values and long-term goals also in the presence of those negative experiences.

The specific research questions are:

* Can the psychological treatment rationale with its focus on psychoeducation, validation, exposure, and acceptance among other therapeutic techniques, preserve cognitive status, increase life satisfaction, improve psychological health, show positive biological changes in individuals with SCD/MCI?
* Are potential treatment effects maintained longitudinally?
* Can significant treatment predictors be identified on treatment outcome?
* How does the participants perceive the treatment?

Hypotheses Main hypothesis

1. The main hypothesis declares that participants obtaining PIPCI will increase their psychological flexibility (AAQ2) compared to participants in the control groups and that this effect will be retained at 6 months follow-up.

Secondary hypotheses

1. The secondary hypotheses declares that participants obtaining PIPCI will improve psychological health (stress measures, quality of life, depression and general health), in correspondence with biomarker changes compared to the control groups
2. An additional secondary hypothesis declares that participants obtaining PIPCI, and participants in the active control group, will improve on the cognitive test measures compared to the waiting list group. However, we do not have any directed hypothesis comparing PIPCI and the active control group.

Exploratory research questions (without any directed hypotheses)

1. Can we identify significant pre-intervention predictors for intervention outcomes?
2. How do participants perceive the intervention?

Methods

Patients will be recruited from the Cognitive Centers at the Karolinska University Hospital, Solna, and Huddinge within Stockholm metropolitan area, where they partake in cognitive examination (i.e., neuropsychological assessments, anamnesis, biological markers etc.). These patients will be younger than 70 years and will have received a diagnosis of SCD or MCI.

Randomization

The identified patients receive verbal and written information about the project. In the next step, patients that express interest for the project signs an informed consent and will then be evaluated in a semi-structured interview, conducted by a psychologist at the Unit of Behavioral Medicine at Karolinska University Hospital, Stockholm, Sweden. Patients that fulfill the inclusion criteria and considered suitable for treatment, are randomized. For the randomization process, the investigators will engage the Karolinska Trial Alliance, Stockholm, Sweden (https://karolinskatrialalliance.se/en/), that is a professional clinical research center at Karolinska University Hospital.

RCT design and groups

One group will receive psychological treatment (experimental group), one group will get cognitive training (active control group), and one group will get the gold standard treatment, which is health information (TAU). After the finalization of the post-intervention evaluations, the TAU group will be randomized to participate in one of the active interventions. Participants need to be present for at least 75 % of the intervention and completed at least 75 % of the homework to be considered adherent. All evaluation assessments will be conducted by blinded assessors. Participants cannot be blinded to their group assignment, which is typical of non-pharmacological intervention trials.

Power calculation

Sample size was calculated with the R package SIMR, which allows power calculations of Linear Mixed Models (LMM). The sample size estimate is based on changes in our primary outcome, AAQ2. The model included the interaction of time (pre- versus post-test 1; continuous) and group (experimental versus active control; factor). The model also had subject ID (factor) as a random effect to account for repeated measurements. The analysis showed that to get a significant difference between the experimental group and the active control group we need at least 40 participants (to have 93% power) in each group. We expect a 15% attrition rate, so an initial recruitment of 120 participants should ensure that about 105 participants remain in the final sample.

Ethical considerations

The project has an approved ethical application (Dnr. 2022-06139-01) by the Regional Ethical Committee in Stockholm and follows the Declaration of Helsinki. Cognitive impairments are often related to progressive decline in cognitive and intellectual abilities. Thus, there is a risk that patients may progress in their decline during the period in which they are included. The investigators therefore need to be watchful on potential progression, and referral to other health care units can be needed if the patient's conditions are changing to the worse. The treatment/rehabilitation might in some cases be perceived as psychologically tough when it comes to behavioral changes. This is not unique for the current study, but often a part of any psychological clinical treatment/rehabilitation. To provide qualified support to the patients, only professional clinicians will interact with the participants. Most of them will be licensed and sanctioned by the Social Board of Health and Welfare (Socialstyrelsen) who is governed by ethical guidelines and the need to protect the patients and their personal information.

Statistical analysis

The continuous longitudinal data derived from the RCT will be analyzed using appropriate growth models (e.g., LMM) that in addition to studying change at the group level also can: model change on the individual level; flexibly incorporate time-varying predictors; handle dependency for repeated observations and provide correct estimates with missing data under largely unconstrained missing data conditions. As a default strategy we will use LMM to analyze the condition by time interaction and will follow established recommendations for model specification and reporting results. In the main analysis, we will compare intervention change between the PIPCI group and the active control group. However, we will also compare the PIPCI group and the active control group with the waiting list group. An alpha level of 0.05 and a 95% CI will be used to evaluate the main and secondary analyses.

In addition to using the growth model framework to investigate predictors of intervention outcomes, we will also apply non-linear models using machine learning methodology, such as support vector machines (SVMs). The SVM fits the separating hyperplane with support from the cases that lie closest to each other in hyperspace but which are of different labels, the support vectors. The developed risk models will mainly predict cognitive test measures (neuropsychological assessments), and biological markers (visual ratings derived from magnetic resonance imaging, and cerebrospinal fluid dementia measures.

The qualitative approach will be conducted in line with consolidated criteria for reporting qualitative research (COREQ), with the aim to examine in-depth participant's experiences of participation in the RCT. Interviews will be conducted with participants in the study after the long-term follow-up. Interviews will be digitally recorded and transcribed, and content analysis will be used in the analysis.

ELIGIBILITY:
* Criteria's for inclusion
* < 75 years.
* SCD or MCI diagnosis. All cognitive MCI-subtypes are eligible.
* Mild to moderate psychological symptoms that are indicated to be related to the patient's CI. The psychological symptoms should affect the patients daily living and behavior, exemplified by avoidance behavior, social anxiety and perceived stigmatization.
* Fluency in the Swedish language.
* The patients should have access to a mobile telephone to be able to receive reminders via Short Message Service (SMS).
* Signed informed consent.
* Criteria's for exclusion
* Dementia diagnosis and/or occurrence of serious illness and/or injury that requires immediate investigation or treatment of another type, or which is expected to worsen in the coming year (i.e., not including dementia)
* Severe psychiatric comorbidity (e.g., high suicide risk), and/or severe psychiatric disorder. This will be assessed in the MINI evaluation and during the clinical cognitive examination).
* Anti-depressant medication introduced or alterations in dosage < 6 months ago (i.e., un-stable dose).
* Mini Mental State Examination (MMSE) score < 26 and/or a Montreal Cognitive Assessment (MoCA) score < 24.
* Stroke or head trauma < 6 months ago.
* Substance abuse

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in psychological flexibility measured with the Acceptance and action questionnaire (AAQ2) | Measurement 1: 1 week prior to the intervention. Measurement 2: Change in AAQ2 from pre-intervention at 1 week post-intervention. Measurement 3: Change in AAQ2 from 1 week post-intervention at 6-month post intervention.
  A psychological health measure (questionaire) measuring the ability to notice and accept interfering thoughts, emotions and bodily sensations without acting on them, to facilitate behaving in accordance with personal values and long-term goals also in the presence of those negative experiences. Scores: 0-49 A low score indicate a more positive outcome.

SECONDARY OUTCOMES:
Change in perceived stress scale (PSS) | Measurement 1: 1 week prior to the intervention. Measurement 2: Change in PSS from pre-intervention at 1 week post-intervention. Measurement 3: Change in PSS from 1 week post-intervention at 6-month post intervention.
  Questionnaire measuring stress related symptoms. Scale: 0-40. A low score indicate a more positive outcome.
Change in Becks Depression Inventory (BDI) | Measurement 1: 1 week prior to the intervention. Measurement 2: Change in BDI from pre-intervention at 1 week post-intervention. Measurement 3: Change in BDI from 1 week post-intervention at 6-month post intervention.
  Questionnaire measuring Depression. Scale_ 0-63. A low score indicate a more positive outcome.
Change in Brunnsvikens Brief Quality of Life Scale (BBQ) | Measurement 1: 1 week prior to the intervention. Measurement 2: Change in BBQ from pre-intervention at 1 week post-intervention. Measurement 3: Change in BBQ from 1 week post-intervention at 6-month post intervention.
  Questionnaire measuring quality of life. Scale: 0-48. A high score indicate a more positive outcome.
Change in Short Form Health Survey (SF-36) | Measurement 1: 1 week prior to the intervention. Measurement 2: Change in SF-36 from pre-intervention at 1 week post-intervention. Measurement 3: Change in SF-36 from 1 week post-intervention at 6-month post intervention.
  Health survey. Scale: Scale: Consist of eight scales that are transformed to 0-100 scales. Lower scores indicate higher disability.
Change in Generalized Anxiety Disorder 7-item Scale (GAD-7) | Measurement 1: 1 week prior to the intervention. Measurement 2: Change from pre-intervention at 1 week post-intervention. Measurement 3: Change from 1 week post-intervention at 6-month post intervention.
  Anxiety estimate. Scale 0-3. A low score indicate a more positive outcome.
Childhood Trauma Questionnaire (CTQ) | Measurement 1: 1 week prior to the intervention. This questionnaire will be evaluated in respect of predicting treatment outcome.
  Questionnaire to identify and measure the prevalence of retrospective childhood trauma. A low score indicate a more positive outcome. Total score is 140, and a low score indicate a more positive outcome.
Client Satisfaction Questionnaire (CSQ-8) | Measurement 1: 1 week post-intervention. Measurement 2: Change from 1 week post-intervention at 6-month post intervention.
  A global measure of client satisfaction with the intervention. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Change in Brief Visuospatial Memory Test Revised (BVMT-R) | Measurement 1: 1 week prior to the intervention. Measurement 2: Change in BVMT-R from pre-intervention at 1 week post-intervention. Measurement 3: Change in BVMT-R from 1 week post-intervention at 6-month post intervention.
  Measuring non-verbal episodic memory. Measured in correct answer. A high score indicate a better performance.
Change in computer-based AX-Continuous Performance Task (CPT) | Measurement 1: 1 week prior to the intervention. Measurement 2: Change in AX-CPT from pre-intervention at 1 week post-intervention. Measurement 3: Change in AX-CPT from 1 week post-intervention at 6-month post intervention.
  Measuring executive functions. Measured in correct answers. A high score (correct answers) and fast response times indicate a good performance.
Change in computer-based reaction time test from Deary-Liewald | Measurement 1: 1 week prior to the intervention. Measurement 2: Change in Deary-Liewald from pre-intervention at 1 week post-intervention. Measurement 3: Change in Deary-Liewald from 1 week post-intervention at 6-month post intervention.
  Measuring reaction times. Measured in correct answers. A high score indicate a good performance.
Change in Design fluency test, D-KEFS | Measurement 1: 1 week prior to the intervention. Measurement 2: Change from pre-intervention at 1 week post-intervention. Measurement 3: Change from 1 week post-intervention at 6-month post intervention.
  Measure aspects of executive functions. Measured in correct answers. A high score (correct answers) and fast response times indicate a good performance.
Change in the computer-based Flanker task | Measurement 1: 1 week prior to the intervention. Measurement 2: Change from pre-intervention at 1 week post-intervention. Measurement 3: Change from 1 week post-intervention at 6-month post intervention.
  Measure aspects of executive functions such as inhibition. Measured in correct answers. A high score (correct answers) and fast response times indicate a good performance.
Change in the computer-based Visual Short-Term Memory Binding Test (VSTMBT) | Measurement 1: 1 week prior to the intervention. Measurement 2: Change from pre-intervention at 1 week post-intervention. Measurement 3: Change from 1 week post-intervention at 6-month post intervention.
  Involves, in the short-time perspective, the ability to hold information in memory especially the integration between surface features, such as shapes and colours
Change in brain derived neuro-tropic factor (BDNF) | Measurement 1: 1 week prior to the intervention. Measurement 2: Change from pre-intervention at 1 week post-intervention. Measurement 3: Change from 1 week post-intervention at 6-month post intervention.
  A biological blood measure, measuring cellular health. Increased activity indicate an increased cellular activity, and a positive outcome.
Change in Interleukin 6 | Measurement 1: 1 week prior to the intervention. Measurement 2: Change from pre-intervention at 1 week post-intervention. Measurement 3: Change from 1 week post-intervention at 6-month post intervention.
  A biological blood measure. Increased interleukin-6 level may be an independent risk factor for disease severity. Thus, we expect lowered levels as a consequence of the interventions.
Change in Hemoglobin HbA1C | Measurement 1: 1 week prior to the intervention. Measurement 2: Change from pre-intervention at 1 week post-intervention. Measurement 3: Change from 1 week post-intervention at 6-month post intervention.
  A blood measure that shows the average blood sugar (glucose) level over the past two to three months. Increased HbA1C level may be an independent risk factor for disease severity. Thus, we expect lowered levels as a consequence of the interventions.
Change in Cortisol | Measurement 1: 1 week prior to the intervention. Measurement 2: Change from pre-intervention at 1 week post-intervention. Measurement 3: Change from 1 week post-intervention at 6-month post intervention.
  A hormone made by the adrenal glands. It helps the body respond to stress etc. Increased Cortisol level may be an independent risk factor for disease severity. Thus, we expect lowered levels as a consequence of the interventions.
Change in C-peptide | Measurement 1: 1 week prior to the intervention. Measurement 2: Change from pre-intervention at 1 week post-intervention. Measurement 3: Change from 1 week post-intervention at 6-month post intervention.
  A measure of pancreatic beta cell function. C-peptide has previously been shown to be negatively correlated with depression level. Thus, we expect than increased C-peptide levels as a consequence of the interventions.
Change in Insulin | Measurement 1: 1 week prior to the intervention. Measurement 2: Change from pre-intervention at 1 week post-intervention. Measurement 3: Change from 1 week post-intervention at 6-month post intervention.
  A hormone that regulates the level of sugar (glucose) in the blood. Previous results indicate that there can be a link between blood sugar dysregulation and mood disorders. We expect increased insulin levels as a consequence of the interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Miia Kivipelto, Professor, Study Director — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wallin A, Kettunen P, Johansson PM, Jonsdottir IH, Nilsson C, Nilsson M, Eckerstrom M, Nordlund A, Nyberg L, Sunnerhagen KS, Svensson J, Terzis B, Wahlund LO, Georg Kuhn H. Cognitive medicine - a new approach in health care science. BMC Psychiatry. 2018 Feb 8;18(1):42. doi: 10.1186/s12888-018-1615-0. PMID 29422020
- [Background] Jessen F, Wolfsgruber S, Wiese B, Bickel H, Mosch E, Kaduszkiewicz H, Pentzek M, Riedel-Heller SG, Luck T, Fuchs A, Weyerer S, Werle J, van den Bussche H, Scherer M, Maier W, Wagner M; German Study on Aging, Cognition and Dementia in Primary Care Patients. AD dementia risk in late MCI, in early MCI, and in subjective memory impairment. Alzheimers Dement. 2014 Jan;10(1):76-83. doi: 10.1016/j.jalz.2012.09.017. Epub 2013 Jan 30. PMID 23375567
- [Background] Winblad B, Palmer K, Kivipelto M, Jelic V, Fratiglioni L, Wahlund LO, Nordberg A, Backman L, Albert M, Almkvist O, Arai H, Basun H, Blennow K, de Leon M, DeCarli C, Erkinjuntti T, Giacobini E, Graff C, Hardy J, Jack C, Jorm A, Ritchie K, van Duijn C, Visser P, Petersen RC. Mild cognitive impairment--beyond controversies, towards a consensus: report of the International Working Group on Mild Cognitive Impairment. J Intern Med. 2004 Sep;256(3):240-6. doi: 10.1111/j.1365-2796.2004.01380.x. PMID 15324367
- [Background] Wicksell RK, Olsson GL, Hayes SC. Psychological flexibility as a mediator of improvement in Acceptance and Commitment Therapy for patients with chronic pain following whiplash. Eur J Pain. 2010 Nov;14(10):1059.e1-1059.e11. doi: 10.1016/j.ejpain.2010.05.001. Epub 2010 Jun 9. PMID 20538493
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724
- [Derived] Ekman U, Kemani MK, Wallert J, Wicksell RK, Holmstrom L, Ngandu T, Rennie A, Akenine U, Westman E, Kivipelto M. Evaluation of a Novel Psychological Intervention Tailored for Patients With Early Cognitive Impairment (PIPCI): Study Protocol of a Randomized Controlled Trial. Front Psychol. 2020 Dec 23;11:600841. doi: 10.3389/fpsyg.2020.600841. eCollection 2020. PMID 33424715